CLINICAL TRIAL: NCT00982150
Title: A Multinational, Multicenter, Open Label Phase to Assess Tolerability and Safety of Talampanel 50mg Tid in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Extension Study of Talampanel for Amyotrophic Lateral Sclerosis (ALS)
Acronym: ALSTAR OL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Core study unsuccessful
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALS-TAL-201-OL
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Talampanel; Open-Label Study; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — talampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Talampanel (Experimental): Talampanel 50mg tid
  Interventions: Drug: Talampanel

INTERVENTIONS:
Drug: Talampanel — 50mg capsules tid

SUMMARY:
This will be an open label treatment extension phase in patients with ALS who have previously participated in the double blind, placebo-controlled ALS-TAL-201 study. This study will make talampanel treatment available to all subjects who completed the double blind placebo-controlled phase of ALS-TAL-201 study and where the investigator and patient consider it to be in the patient's interest to receive talampanel 50mg three times daily (tid). It will also enable the exploration of long-term safety and tolerability of talampanel 50mg tid.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed 52 weeks of treatment of the double blind placebo-controlled phase of ALS-TAL-201.
* Women must be postmenopausal, surgically sterile, or using adequate birth control methods.
* Patients must be willing and able to give written informed consent prior to performing any open-label study procedures.

Exclusion Criteria:

* Patients with ECG signs of Brugada syndrome and/ or complete or incomplete Right Bundle Branch Block
* Patients using any of the following:

  * Chronic use of lithium carbonate
  * Chronic use of mecasermin (rhIGF-1)
  * Chronic use of minocycline
  * Chronic use of more than 600mg/day coenzyme Q10
  * Chronic use of any marketed drug, if its use was not clearly indicated for any underlying medical condition other than ALS (symptomatic drugs for ALS and supplements allowed)
* Patients participating in any other investigational drug study and use of any other investigational drug
* Patients taking drugs that may interact with Talampanel
* Females who are pregnant or nursing.
* Females of child-bearing potential who do not practice medically acceptable methods of contraception.
* Any condition of the patient which the investigator feels may interfere with participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
ALSFRS-R | every 4 weeks

SECONDARY OUTCOMES:
Vital Signs, ECG, Adverse Event Reports | every 26 weeks